CLINICAL TRIAL: NCT06359197
Title: Feasibility Study for Investigating the Effect of Caffeine Consumption on Protein Biomarkers Related to Cardiovascular Disease
Brief Title: Effect of Caffeine Consumption on Protein Biomarkers and Cardiovascular Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024-17022-GRA
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Caffeine; Protein Biomarkers; Proteomics; Feasibility; TASSO; Dried Blood Spot (DBS); Capillary blood
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: An external party will prepare an equal number of kits (n=18) containing all the required materials for the participants, both in the placebo and caffeine group. They will assign a unique random number to each of the packages; each number will correlate to either the placebo or caffeine group. When a participant agrees to the study, they will be given a unique participant ID number ranging from 0-36. Then, the external party will use a random number generator to pick the kit given to that participant. They will record the number associated with that kit, and link the kit number to the participant ID for tracking purposes. At the end of the study, the investigators will determine which participants received caffeine vs placebo based on the assigned random numbers.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Caffeine - Phase 1 (Experimental): The sample size of this arm is 5 participants. In this arm, participants will have to come to the Population Health Research Institute building to complete study procedures. They will undergo an overnight fast of at least 8 hours, then undergo blood collection by intravenous sampling, as well as by the TASSO+ device and finger prick and collection on Whatman Protein 903 Saver Cards. They will then ingest a 400mg dose of caffeine and remain fasted for the following 6 hours. At 3 hours and 6 hours post caffeine consumption, participants will have their blood collected in the same manner as the initial blood collection.
  Interventions: Drug: Caffeine Pill; Device: TASSO+ Device; Device: Finger prick and collection on Whatman Protein 903 Saver Cards; Device: Intravenous Sampling
- Control - Phase 1 (Placebo Comparator): The sample size of this arm is 5 participants. In this arm, participants will have to come to the Population Health Research Institute building to complete study procedures. They will undergo an overnight fast of at least 8 hours, then undergo blood collection by intravenous sampling, as well as by the TASSO+ device and finger prick and collection on Whatman Protein 903 Saver Cards. They will then ingest 2 placebo pills and remain fasted for the following 6 hours. At 3 hours and 6 hours post caffeine consumption, participants will have their blood collected in the same manner as the initial blood collection.
  Interventions: Drug: Placebo; Device: TASSO+ Device; Device: Finger prick and collection on Whatman Protein 903 Saver Cards; Device: Intravenous Sampling
- Caffeine - Phase 2 (Experimental): The sample size of this arm is 13 participants. In this arm, participants will remain at home to complete study procedures. They will undergo an overnight fast of at least 8 hours, then self-collect blood using the TASSO+ device. They will then ingest a 400mg dose of caffeine and remain fasted for the following 6 hours. At 3 hours and 6 hours post caffeine consumption, participants will collect their blood using the TASSO+ device.
  Interventions: Drug: Caffeine Pill; Device: TASSO+ Device
- Control - Phase 2 (Placebo Comparator): The sample size of this arm is 13 participants. In this arm, participants will remain at home to complete study procedures. They will undergo an overnight fast of at least 8 hours, then self-collect blood using the TASSO+ device. They will then ingest 2 placebo pills and remain fasted for the following 6 hours. At 3 hours and 6 hours post caffeine consumption, participants will collect their blood using the TASSO+ device.
  Interventions: Drug: Placebo; Device: TASSO+ Device

INTERVENTIONS:
Drug: Caffeine Pill — Participants would take two Wake-Ups 200mg Caffeine tablets to meet the target dose of 400mg of caffeine. These are a registered natural health product with Health Canada (NPN 80003474). They are developed by Adrem Brands, which was established in 1951. Quality control testing is performed at a third-party independent lab, Nucro-Technics, which is audited by Health Canada and the US FDA. This ensures that the caffeine tablets comply with Health Canada standards. The tablets contain caffeine anhydrous-a processed, dehydrated form of caffeine-which allows for a standard dose per tablet. The tablets are sugar-free, which reduces the confounding effect of sugar on our results; thus, the investigators can be more confident that the obtained results are reflective of the association between caffeine and the CVD-related protein biomarkers.
  Arms: Caffeine - Phase 1; Caffeine - Phase 2
Drug: Placebo — Participants would take two placebo pills to match the dosage of the intervention group. The investigators will use empty vegetable capsules from Health Bloom as the placebo for the control group. These capsules contain no contaminants or additives and are free from the common allergens. They are sugar-free-unlike most placebo pills, which reduces the confounding effect of sugar on our results. They are developed by Health Bloom, which is a Canadian company established in 2015. These capsules undergo testing at various stages of production to ensure purity and quality control. Each ingredient is tested prior to formulation, and the final capsules are subjected to thorough testing post-development. The capsules are white, and similar in appearance to the caffeine pill given to participants in the intervention group.
  Arms: Control - Phase 1; Control - Phase 2
Device: TASSO+ Device — TASSO+ is a blood lancet device that uses negative pressure to draw capillary blood from the upper arm into a standard SST tube of volume 500μL. The small volume of blood collected makes this device less invasive than traditional collection methods. It is also safer and easier to use since it offers automated sample collection. TASSO manufactures a number of special devices for capillary blood sampling that have been validated as safe for consumer use, and the Tasso+ device is licensed with Health Canada for research use.
Device: Finger prick and collection on Whatman Protein 903 Saver Cards — The Whatman Protein 903 Saver Card is a specialized filter paper designed for the collection, storage, and elution of biological samples, including blood. It contains five half-inch circles that hold 75 to 80 µL of blood, making it an efficient and reliable method of obtaining dried blood spot (DBS) samples. The participant's finger will be pricked using a sterile, disposable lancet, and drops of blood will be collected on the Whatman 903 Protein Saver Card to fill nine ½ inch discs via capillary action. The blood spots will be allowed to dry at ambient temperature (21°C) for two hours. Whatman Protein 903 Saver Cards undergo strict quality control and GMP manufacturing standards, which ensures high quality and reproducibility.
  Arms: Caffeine - Phase 1; Control - Phase 1
Device: Intravenous Sampling — Blood will be collected from the medial cubital vein according to the standard venous blood sampling protocol into an EDTA tube with a volume up to 4mL.
  Arms: Caffeine - Phase 1; Control - Phase 1

SUMMARY:
Caffeine is one of the most widely consumed substances worldwide. This study looks to test and measure the changes in different biomarkers in the blood before and after having caffeine using capillary and venous blood sampling methods. A biomarker is a measurable indicator of biological processes. The primary goal of this clinical trial is to evaluate participant rate and adherence. It will also learn about how caffeine affects different biomarkers that may be related to cardiovascular disease. Finally, it will assess the accuracy of the capillary blood samples compared to the venous blood samples. The main questions it aims to answer are:

* What is the feasibility of recruiting and retaining participants?
* Are the study procedures appropriate to be translated to a larger future study?

Researchers will compare caffeine to a placebo (a look-alike substance that contains no drug) to see if

Participants will:

* Be randomly assigned to the control group or the caffeine group. Individuals in the control group will be taking a placebo pill with no effect and those in the caffeine group will be taking 400mg of caffeine in pill form.
* Be asked to undergo a fast of at least 8 hours overnight before taking two placebo pills or the 400 mg of caffeine via two caffeine pills. They will be required to stay fasted for 6 hours after taking the pill as well. The total time fasted will be at least 14 hours.
* Have blood collected using three different methods before taking the two pills, 3 hours after taking the pills and 6 hours after taking the pills. The 3 methods include intravenous (IV) blood sampling, finger prick and collection on Whatman 903 Protein Saver Card and collection using the TASSO+ device. The TASSO+ blood collection device is a small capillary blood collection device that is designed to be easy to use and able to be used outside of a hospital/lab setting. Whatman 903 Protein Saver Cards are special filter paper with five circles for samples, that are designed for the collection and storage of blood.

DETAILED DESCRIPTION:
Proteomic biomarkers related to disease risk factors may shed light on the pathogenesis of different diseases. There is a knowledge gap in the effects of lifestyle interventions on the proteome, mainly because collection of blood samples by venipuncture for proteomics analysis is tedious and expensive. Discovering an at-home capillary blood collection method with samples that contain protein profiles that mirror or can be correlated to those of venous samples has the potential to greatly improve access to research studies. Cardiovascular diseases (CVD) are the most common cause of death worldwide. Caffeine is a commonly consumed substance. Many studies have shown a relationship between caffeine and reduced risk of CVD; however, the mechanisms remain mostly unknown.

The investigators are conducting a two-part feasibility study examining the effect of caffeine consumption on the relative levels of 92 cardiovascular-related protein biomarkers in samples obtained using different blood collection technologies to compare protein profiles between capillary and venous blood samples and further clarify the protective mechanisms of caffeine in mitigating CVD risk. By integrating both of these components into a single trial, the investigators aim to reduce the burden placed on participants, making the study easier and more accessible.

For the preliminary testing of the at-home blood collection methods compared with intravenous sampling, a group of 10 individuals (evenly split between male and female) will be recruited. In this phase, participants will be subject to blood collection by intravenous sampling, as well as the TASSO+ device and finger prick and collection on Whatman Protein 903 Saver Cards. After the first portion of the study is complete, data from the 10 patients will be analyzed to determine the most accurate and reliable capillary blood collection device. This sampling device will show a reasonable correlation to venipuncture, with a threshold of correlation above 70%.

For the larger at-home testing of the selected blood collection method, a group of 26 individuals will participate, again, with an even split between males and females. Participants in this second cohort will no longer have to come on premise for intravenous sampling. They can complete the entire study remotely, further reducing logistical challenges. In this phase, blood will only be collected using the capillary blood collection device that best correlates with venipuncture as validated in the first part of the study.

After the second portion of the study is complete, data from the first 10 participants will be integrated and compared with data from the second 26 participants to evaluate the effect of caffeine vs placebo on biomarkers, as well as identify any significant differences between the two cohorts.

In both phases, participants will undergo a fast of at least 8 hours prior to the administration of the caffeine or placebo. Following this fast, blood will be collected (either at home or in the lab) prior to the ingestion of the caffeine pill or placebo. Blood will also be collected at 3 and 6 hours after the ingestion of the caffeine pill or placebo. Blood samples will either be collected in the lab or collected at-home then mailed back to the lab, and stored in a -80°C freezer until proteomic analysis may be conducted to investigate the changes in biomarkers.

With this being a feasibility study, the investigators are hoping to see some results from this sample size, then translate their findings to a larger study with more participants conducted over a longer period of time in the future.

ELIGIBILITY:
Inclusion Criteria:

- Participants must be over the age of 18 to participate in the study. This is based on 400mg of caffeine being deemed safe for healthy adults.

Exclusion Criteria:

* Participants are not to be pregnant or trying to get pregnant or lactating as the recommended caffeine consumption for these individuals is less than what would be administered in this study.
* Individuals who are diabetic will be excluded from this study due to the fasting period, potentially leading to a low blood sugar state.
* Individuals with the following conditions will be excluded from the study: Hypertension or a history of hypertension Glaucoma Thyroid disease Heart disease Seizure disorder The investigators will screen the participant's medical conditions and not include anyone whose condition may interfere.
* Individuals who experience anxiety or have been diagnosed with other mental illnesses will want to consider their participation in this study. Those who experience anxiety may experience more anxiety-related symptoms with the consumption of caffeine. The investigators will screen participant's for anxiety-related disorders.
* Individuals who have recently undergone major surgery. Major surgery is any intervention that has resulted in the penetration and opening of a body cavity (i.e., chest or abdominal). Recent is within the last month.
* Individuals who are taking medication which may have adverse interactions with caffeine will be excluded from the study. The investigators will screen the participant's medications and not include anyone whose medications may interfere.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2024-08-10 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Participant rate | From enrollment to the end of intervention at 6 hours post caffeine or placebo consumption
  To evaluate participant rate, the investigators will determine (1) how many participants enter the study at a time, (2) how long it takes to recruit enough participants into the study, and (3) what are the refusal rates for participation. Their goal is to have a participant rate of 75%, meaning that they are able to recruit 75% of the people that are approached.
Participant Adherence | From enrollment to the end of intervention at 6 hours post caffeine or placebo consumption
  To evaluate participant adherence, the investigators will determine the retention and follow-up rates as the participants move through the study. Their goal is to have an adherence rate of 95% as this will help to avoid attrition bias, which will ensure that there will be no significant differences between the analyzed cohort vs. participants who were lost to follow-up or withdrew from the study.
Participant satisfaction | From enrollment to the end of intervention at 6 hours post caffeine or placebo consumption
  User experience with the capillary blood collection devices will be evaluated using a satisfaction survey. Participants will rate their experience using a 5-point Likert scale ranging from extremely difficult (1 point) to extremely easy (5 points) for four questions related to ease-of-use, and from not usable (1 point) to no pain (5 points) for one question related to comfort of use. The investigators will consider a score of ≥20 to indicate acceptability and suitability of the device. They will consider achieving a satisfaction score of ≥20 from >80% of participants to be feasible.

SECONDARY OUTCOMES:
Significant changes in biomarkers observed after the ingestion of caffeine | From enrollment to the end of intervention at 6 hours post caffeine or placebo consumption
  The investigators plan to investigate the effect of caffeine consumption on the relative levels of 92 protein biomarkers included in the OLINK CVD III panel. This will shed light on specific proteins and pathways that underpin caffeine's potential protective role against CVD. This will provide a more comprehensive understanding of the mechanisms involved in caffeine's influence on CVD risk. The protein biomarkers expressed in the samples will be measured using OLINK proteomic analysis which will produce an NPX value for each of the measured biomarkers on the panels being used with the collected blood samples. They will compare the biomarker levels at the different timepoints post-caffeine consumption to those at baseline (timepoint 0).
Determine the correlation between capillary sampling and intravenous sampling | From enrollment to the end of intervention at 6 hours post caffeine or placebo consumption in phase 1 cohort
  To accomplish this objective, the investigators need to determine how well the protein biomarker levels correlate between the samples collected from the different capillary microsampling devices (TASSO+ device and finger prick and collection on Whatman Protein 903 Saver Cards) and intravenous blood sampling.
Determine the stability of capillary samples | From enrollment to the end of intervention at 6 hours post caffeine or placebo consumption
  The investigators need to determine the relative stability of the protein biomarkers measured from the different sample types under different, week-long preanalytical storage conditions (-80 C, 20°C, and 37°C for 7 days). These conditions mimic possible temperature fluctuations during the shipping chain of the remote samples from the end-user to the lab.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Pare, MD, Principal Investigator — Population Health Research Institute
Locations (3):
- Canada (3):
  - David Braley Research Institute, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University, Department of Pathology and Molecular Medicine, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Jett JD, Beck R, Tyutyunnyk D, Sanchez J, Lopez-Cruzan M, Ginsburg BC, McPherson SM, Javors MA, McDonell MG, Hill-Kapturczak N. Validation of the quantification of phosphatidylethanol 16:0/18:1 concentrations in TASSO-M20 devices. Alcohol Clin Exp Res (Hoboken). 2023 Apr;47(4):748-755. doi: 10.1111/acer.15024. Epub 2023 Feb 21. PMID 36811188
- [Background] Shen X, Kellogg R, Panyard DJ, Bararpour N, Castillo KE, Lee-McMullen B, Delfarah A, Ubellacker J, Ahadi S, Rosenberg-Hasson Y, Ganz A, Contrepois K, Michael B, Simms I, Wang C, Hornburg D, Snyder MP. Multi-omics microsampling for the profiling of lifestyle-associated changes in health. Nat Biomed Eng. 2024 Jan;8(1):11-29. doi: 10.1038/s41551-022-00999-8. Epub 2023 Jan 19. PMID 36658343
- [Background] Numao S, Uchida R, Kurosaki T, Nakagaichi M. Differences in circulating fatty acid-binding protein 4 concentration in the venous and capillary blood immediately after acute exercise. J Physiol Anthropol. 2021 Feb 10;40(1):5. doi: 10.1186/s40101-021-00255-z. PMID 33568227
- [Background] Wik L, Nordberg N, Broberg J, Bjorkesten J, Assarsson E, Henriksson S, Grundberg I, Pettersson E, Westerberg C, Liljeroth E, Falck A, Lundberg M. Proximity Extension Assay in Combination with Next-Generation Sequencing for High-throughput Proteome-wide Analysis. Mol Cell Proteomics. 2021;20:100168. doi: 10.1016/j.mcpro.2021.100168. Epub 2021 Oct 27. PMID 34715355
- [Background] Strimbu K, Tavel JA. What are biomarkers? Curr Opin HIV AIDS. 2010 Nov;5(6):463-6. doi: 10.1097/COH.0b013e32833ed177. PMID 20978388
- [Background] O'Keefe JH, DiNicolantonio JJ, Lavie CJ. Coffee for Cardioprotection and Longevity. Prog Cardiovasc Dis. 2018 May-Jun;61(1):38-42. doi: 10.1016/j.pcad.2018.02.002. Epub 2018 Feb 21. PMID 29474816
- [Background] Brown J, Kreiger N, Darlington GA, Sloan M. Misclassification of exposure: coffee as a surrogate for caffeine intake. Am J Epidemiol. 2001 Apr 15;153(8):815-20. doi: 10.1093/aje/153.8.815. PMID 11296156
- [Background] Lewis M, Bromley K, Sutton CJ, McCray G, Myers HL, Lancaster GA. Determining sample size for progression criteria for pragmatic pilot RCTs: the hypothesis test strikes back! Pilot Feasibility Stud. 2021 Feb 3;7(1):40. doi: 10.1186/s40814-021-00770-x. PMID 33536076
- [Background] Lebeau PF, Byun JH, Platko K, Saliba P, Sguazzin M, MacDonald ME, Pare G, Steinberg GR, Janssen LJ, Igdoura SA, Tarnopolsky MA, Wayne Chen SR, Seidah NG, Magolan J, Austin RC. Caffeine blocks SREBP2-induced hepatic PCSK9 expression to enhance LDLR-mediated cholesterol clearance. Nat Commun. 2022 Feb 9;13(1):770. doi: 10.1038/s41467-022-28240-9. PMID 35140212
- [Background] Temple JL, Bernard C, Lipshultz SE, Czachor JD, Westphal JA, Mestre MA. The Safety of Ingested Caffeine: A Comprehensive Review. Front Psychiatry. 2017 May 26;8:80. doi: 10.3389/fpsyt.2017.00080. eCollection 2017. PMID 28603504
- [Background] Nawrot P, Jordan S, Eastwood J, Rotstein J, Hugenholtz A, Feeley M. Effects of caffeine on human health. Food Addit Contam. 2003 Jan;20(1):1-30. doi: 10.1080/0265203021000007840. PMID 12519715
- [Background] Eshghi A, Pistawka AJ, Liu J, Chen M, Sinclair NJT, Hardie DB, Elliott M, Chen L, Newman R, Mohammed Y, Borchers CH. Concentration Determination of >200 Proteins in Dried Blood Spots for Biomarker Discovery and Validation. Mol Cell Proteomics. 2020 Mar;19(3):540-553. doi: 10.1074/mcp.TIR119.001820. Epub 2020 Jan 2. PMID 31896676
- [Background] Bjorkesten J, Enroth S, Shen Q, Wik L, Hougaard DM, Cohen AS, Sorensen L, Giedraitis V, Ingelsson M, Larsson A, Kamali-Moghaddam M, Landegren U. Stability of Proteins in Dried Blood Spot Biobanks. Mol Cell Proteomics. 2017 Jul;16(7):1286-1296. doi: 10.1074/mcp.RA117.000015. Epub 2017 May 13. PMID 28501802
- [Background] Fontaine E, Saez C. Capillary blood stability and analytical accuracy of 12 analytes stored in Microtainers(R). Pract Lab Med. 2023 Jul 5;36:e00325. doi: 10.1016/j.plabm.2023.e00325. eCollection 2023 Aug. PMID 37649539
- [Background] Knitza J, Tascilar K, Vuillerme N, Eimer E, Matusewicz P, Corte G, Schuster L, Aubourg T, Bendzuck G, Korinth M, Elling-Audersch C, Kleyer A, Boeltz S, Hueber AJ, Kronke G, Schett G, Simon D. Accuracy and tolerability of self-sampling of capillary blood for analysis of inflammation and autoantibodies in rheumatoid arthritis patients-results from a randomized controlled trial. Arthritis Res Ther. 2022 May 25;24(1):125. doi: 10.1186/s13075-022-02809-7. PMID 35614488
- [Background] Wickremsinhe E, Fantana A, Berthier E, Quist BA, Lopez de Castilla D, Fix C, Chan K, Shi J, Walker MG, Kherani JF, Knoderer H, Regev A, Harding JJ. Standard Venipuncture vs a Capillary Blood Collection Device for the Prospective Determination of Abnormal Liver Chemistry. J Appl Lab Med. 2023 May 4;8(3):535-550. doi: 10.1093/jalm/jfac127. PMID 36533519
- [Background] Khiali S, Agabalazadeh A, Sahrai H, Bannazadeh Baghi H, Rahbari Banaeian G, Entezari-Maleki T. Effect of Caffeine Consumption on Cardiovascular Disease: An Updated Review. Pharmaceut Med. 2023 Mar;37(2):139-151. doi: 10.1007/s40290-023-00466-y. Epub 2023 Mar 30. PMID 36995515
- See also: Whatman 903 Protein Saver Cards — https://www.sigmaaldrich.com/CA/en/product/aldrich/wha10534612
- See also: OLINK Target 96 CVD III panel — https://olink.com/products-services/target/cardiometabolic-panel/
- See also: TASSO+ Device — https://www.tassoinc.com/tasso-plus
- See also: Caffeine pills used in study — https://wake-ups.com/products/wake-ups-200mg-caffeine-tablets-3-pack
- See also: Placebo pills used in study — https://healthbloom.ca/collections/empty-vegetable-capsules/products/1000-empty-vegetable-capsules-white-size-0